CLINICAL TRIAL: NCT06512194
Title: An Investigation of Strategies to Understand and Optimize the Antidepressant Effects of Psilocybin (The OPTIMIZE Study)
Brief Title: Investigation to Understand and Optimize Psilocybin
Acronym: OPTIMIZE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Charles Raison (Other)
Collaborators: Usona Institute (Other); Tiny Blue Dot Foundation (Other); Steadman Philippon Research Institute (Other); Emory University (Other)
Responsible Party: Sponsor-Investigator, Charles Raison, Vail Health Behavioral Health Innovation Center Director, Vail Health Behavioral Health
Organization: Vail Health Behavioral Health (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20243954
Record Dates: First submitted 2024-07-16; First posted 2024-07-22 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Depression
Keywords: depression; psilocybin; psychedelics; transcutaneous auricular vagus nerve stimulation; depressive symptoms; well-being; adverse events; ecological momentary assessment; electronically activated recorder; dynamical complexity assessment
MeSH Terms: conditions — Depression | interventions — Psilocybin

STUDY DESIGN:
Intervention Model Description: All subjects will receive a single 25 mg dose of psilocybin administered within a "set and setting" (SaS) framework of psychological support provided by trained clinicians. Post-dosing, subjects will be randomized to 1) taVNS, 2) sham taVNS, or 3) no taVNS.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Group 1: Psilocybin + taVNS (Experimental): Participants in this arm will receive a single 25 mg dose of psilocybin, followed by twice-daily sessions of taVNS for 7 consecutive days. Each taVNS session will be paired with music and prompts related to the participant's psilocybin experience.
  Interventions: Drug: Psilocybin; Device: Transcutaneous Auricular Vagus Nerve Stimulation (taVNS)
- Group 2: Psilocybin + Sham taVNS (Sham Comparator): Participants in this arm will receive a single 25 mg dose of psilocybin, followed by twice-daily sham taVNS sessions for 7 consecutive days. Each sham session will be paired with music and prompts related to the participant's psilocybin experience.
  Interventions: Drug: Psilocybin; Device: Sham taVNS
- Group 3: Psilocybin + No taVNS (Active Comparator): Participants in this arm will receive a single 25 mg dose of psilocybin, followed by no additional intervention. They will receive the standard psychological support related to their psilocybin experience, but no taVNS or sham device will be used.
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — The psilocybin used in this study is synthesized under Good Manufacturing Practice (GMP) guidelines and is provided in a capsule containing 25 mg of synthetic psilocybin.
  Other Names: Psilocybine; Psilocibin; Usona Institute Psilocybin
Device: Transcutaneous Auricular Vagus Nerve Stimulation (taVNS) — Participants will be provided with a taVNS device and trained on its use. The device delivers gentle stimulation to the left ear.
  Other Names: taVNS
  Arms: Group 1: Psilocybin + taVNS
Device: Sham taVNS — Participants will be provided with a taVNS device and trained on its use. The device delivers gentle stimulation to the left ear. In the sham condition, the device will simulate the sensations of active taVNS without delivering therapeutic stimulation.
  Arms: Group 2: Psilocybin + Sham taVNS

SUMMARY:
This study will examine the effects of a single dose of psilocybin, administered with psychological support, on symptoms of depression. It will also assess whether different post-dosing interventions, including a non-invasive technique called transcutaneous auricular Vagus Nerve Stimulation (taVNS), influence various psychological and behavioral outcomes. In addition, the study will explore objective measures of real-world social behavior and identify early behavioral responses that may be associated with long-term treatment outcomes.

DETAILED DESCRIPTION:
One hundred forty-one adults ages 18 to 70 experiencing a major depressive episode of at least 60 days duration of moderate or greater severity at screening will be enrolled to obtain evaluable data on approximately 120 subjects.

All subjects will receive a single 25 mg dose of psilocybin using a "set and setting" therapeutic approach that will include 1) several hours of preparatory sessions prior to dosing and 2) the presence of two facilitators throughout the dosing session; and 3) several post dosing integration sessions with a facilitator.

Following the psilocybin dosing session, subjects will be randomized to 1) taVNS (7 days of twice daily taVNS), 2) sham taVNS (7 days of twice daily sham taVNS), or 3) no taVNS.

Both taVNS and sham sessions will include guided prompts encouraging participants to reflect on key aspects of their psychedelic experience, accompanied by music previously used during the psilocybin dosing session.

Participants will complete assessments at multiple time points to evaluate depression, anxiety, well-being, functional disability, quality of life, social behavior, suicidal ideation, and adverse events before and after psilocybin dosing.

ELIGIBILITY:
Inclusion Criteria:

Current diagnosis of Major Depressive Disorder (MDD), with a depressive episode lasting ≥ 60 consecutive days at the time of screening, as confirmed by structured clinical interview

Medically healthy, as determined by the screening physician, with no significant medical conditions that would interfere with participation or affect the safety of the subject.

Exclusion Criteria:

History or presence of any psychiatric or medical condition that, in the opinion of the investigator, could pose a safety risk, interfere with participation, or confound study results (e.g., bipolar disorder, psychosis, seizure disorder, or cardiovascular disease).

Known family history of a psychotic disorder (e.g., schizophrenia or schizoaffective disorder) in a first-degree relative (biological parent, full sibling, or child).

Current active suicidal ideation with a specific plan within the prior 2 weeks, as assessed via clinical interview and validated instrument (e.g., C-SSRS).

Suicide attempt within the prior 6 months, regardless of intent or lethality.

Current diagnosis of a substance use disorder

Abnormal ECG at screening that may increase risk during participation (e.g., prolonged QTc, arrhythmias, or other clinically significant findings as determined by the study physician).

Unwilling or unable to discontinue prescription psychotropic medications (e.g., antidepressants, antipsychotics, anxiolytics, lithium, anticonvulsants, or mood stabilizers) for the duration of study participation, including any necessary washout period as determined by the investigator.

Any condition, finding, or behavior (including suspected deception or noncompliance) that, in the opinion of the investigator, renders the participant unsuitable for the study or likely to interfere with the integrity of the data or safety of the subject.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Estimated)
Dates: Start 2025-05-13 (Actual); Primary Completion 2029-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Montgomery-Åsberg Depression Rating Scale (MADRS) score | Baseline 2, Week 8 Post-Psilocybin Dosing
  The MADRS is a 10-item depression rating scale that includes questions on the following symptoms: 1. Reported sadness, 2. Apparent sadness, 3. Inner tension, 4. Reduced sleep, 5. Reduced appetite, 6. Concentration difficulties, 7. Lassitude, 8. Inability to feel, 9. Pessimistic thoughts, and 10. Suicidal thoughts. Items are scored via a blinded clinical interview and rated to capture the patient's clinical state over the prior week. Each item yields a score of 0 to 6, and higher scores indicate more severe depression. The overall score ranges from 0 to 60. For this study, the structured MADRS interview will be used.
PROMIS Ability to Participate in Social Roles and Activities - Short Form 8a | Baseline 2, Week 8 Post-Dose
  An 8-item validated measure assessing an individual's perceived ability to engage in social roles and activities, such as work, family responsibilities, and leisure. Participants rate each item on a 5-point Likert scale. Total score can range from 8 to 40 with higher scores indicating greater functional ability and social participation.
Quality of Life Enjoyment and Satisfaction Questionnaire Short-Form (Q-LES-Q) score | Baseline 2, Week 8 Post-Dose
  The Short Form version (Q-LES-Q-SF) will be used in this trial. The measure contains 16 items that assess quality of life. A total score is derived from summing the first 14 items on the scale, with the last 2 items serving as stand-alone queries. Total score can range from 14 to 70 with higher scores indicating better quality of life.

SECONDARY OUTCOMES:
Electronically Activated Recorder (EAR) | Up to 55 days
  The EAR is a naturalistic observation method that uses an audio recording app worn by subjects to silently and unobtrusively record short samples of ambient sounds while subjects go about their daily lives. These recordings can then be transcribed for subjects' natural daily speech, as well as coded for a wide range of aspects of subjects' objectively assessed locations, activities, conversations, social environments, and other behaviors. In the present study, the EAR allows us to measure how subjects' daily behaviors, activities and social interactions change over the course of the study.
Voicediary | Up to 35 days
  Voicediaries will be collected via the Fabla Voicediary App. The app will collect brief speech samples from subjects' talking about (a) the events of their days and (b) retrospective reflections on their experience of psilocybin (after dosing).
Ecological Momentary Assessment (EMA) | Up to 35 days
  EMA will be conducted via the Fabla Voicediary app. The app will send notifications to subjects' smartphones for assessments three times per day. Each item on the assessments will include 2 slider-type items assessing valence and arousal, 3 free response items assessing current context, 2 items assessing connectedness, 1 item assessing sense of meaning, and 2 collaboratively developed items that are personalized to the subject. In addition, one end-of-day assessment will also include 1 item about hours of sleep the previous night, 1 item about substance use in the past 24 hours, and 1 item asking whether subjects have had conversations about their upcoming (during pre-dosing) or past (during post-dosing) psilocybin experiences, and with whom.
Challenging Experiences Questionnaire (CEQ) score | Day 1 Post-Dose, Week 8 Post-Dose
  The CEQ is a 26-item questionnaire that consists of seven factors of challenging experience with psilocybin mushrooms: fear, grief, feeling of losing your sanity (insanity), feel as though you are dying (death), feelings of isolation, physiological distress, and paranoia. The CEQ uses a 6-point response scale [0: None/not at all, 1: So slight cannot decide, 2: Slight, 3: Moderate, 4: Strong; 5: Extreme (more than ever before in my life)] to indicate the degree to which a participant experiences each of a series of subjective effects during their psilocybin session. Total CEQ score is expressed as the percentage of the total possible ratings on the scale. Total score can range from 0-100% with higher scores indicating a greater challenging experience.
Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS) score | Baseline 1, Baseline 2, Week 2 Post-Dose, Week 4 Post-Dose, Week 8 Post-Dose
  The WEMWBS has 14 questions scored using a five-point Likert scale. The items are all worded positively and cover both feeling and functioning aspects of mental wellbeing. Items on the questionnaire are rated on a 5-point scale, where 1= "None of the time", 2= "rarely", 3= "some of the time", 4= "often", 5= "all the time". The scale is scored by summing the response to each item. The minimum scale score is 14 and the maximum is 70. Scores reflect feelings and thoughts in the two weeks prior to answering the questionnaire with higher scores indicating better well-being.
Psychedelic Assisted Therapy Adverse Events (PATAE) | Baseline 1, Baseline 2, Day 1 Post-Dose, Week 1 Post-Dose, Week 2 Post-Dose, Week 4 Post-Dose, Week 8 Post-Dose
  The PATAE was developed to assess pre-dosing and post-acute dosing adverse events that may occur during psychedelic-assisted therapy due to the pharmacologic and psychotherapeutic components, as well as their interaction. The PATAE consists of 54 items that assess across 7 domains: sociocultural, psychospiritual, interpersonal, behavioral, psychotherapy-related, and perceptual.
30-item Mystical Experiences Questionnaire (MEQ30) score | Day 1 Post-Dose, Week 8 Post-Dose
  The MEQ30 is a 30-item self-report measure developed to assess the effects of classic psychedelics in laboratory studies. It covers the major dimensions of the classic mystical experience: unity, transcendence, noetic quality, sacredness, positive mood, and ineffability/paradoxicality. The MEQ has 4 sub scales: 1) transcendence, 2) positive mood, 3) ineffability, and 4) mystical. The total possible range for each sub scale and total score is 0-100% with higher percentages indicating a larger mystical experience. Typically, a complete mystical experience is defined as scoring 60% or more on all four MEQ30 sub scales.
Emotional Breakthrough Inventory (EBI) score | Day 1 Post-Dose, Week 8 Post-Dose
  The EBI is a 6-item self-report scale that assesses the presence and severity of emotionally challenging/distressing experiences that occur during a psychedelic experience. The scale utilizes visual analog responses captured on a line anchored by "not at all" on one end and "very much so" on the other. Experiences queried include 1) facing emotionally difficult feelings that are usually pushed aside; 2) experiencing a resolution of a personal conflict/trauma; 3) being able to explore challenging emotions and memories; 4) having an emotional breakthrough; 5) getting a sense of closure on an emotional problem, and 6) achieving an emotional release followed by a sense of relief. The total possible score ranges from 0-100 with higher scores indicating a greater emotional breakthrough.
Psychological Insight Questionnaire (PIQ) score | Day 1 Post-Dose, Week 8 Post-Dose
  The PIQ is a 23-item instrument designed to query self-perceived attainment of insight during a psychedelic experience. It comprises two subscales: (a) Avoidance and Maladaptive Patterns Insights and Goals; and (b) Adaptive Patterns Insights. Sub scale and total scores range from 0 to 5 with a higher score indicating great psychological insight.
Ego Dissolution Inventory (EDI) score | Day 1 Post-Dose, Week 8 Post-Dose
  The EDI is an 8-item self-report scale designed to measure ego-dissolution. Each item is scored on a visual analogue scale from 0 to 100 with the following statements at the lower and upper end, respectively: "No, not more than usually" and "Yes, I experienced this completely/entirely." The total possible range of scores for the EDI is 0-100 with higher scores indicating a greater ego dissolution.
Awe Experiences Questionnaire - Short Form (AWE-SF) score | Day 1 Post-Dose, Week 8 Post-Dose
  The AWE-SF is a 12-item self-report scale that measures the state of awe. Each items is rated on a scale of 1 to 7, with 1 representing "Strongly Disagree" and 7 representing "Strongly Agree". The total possible range of scores for the AWE is 12-84 with higher scores indicating a greater awe.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Raison, MD, Principal Investigator — Vail Health Behavioral Health
Locations (1):
- Vail Health Behavioral Health, Edwards, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data including, but not limited to, demographics, questionnaires, and adverse events will be made available upon request.
Time Frame: Following publication of primary study findings.
Access Criteria: EAR/ Voicediary/ EMA Data: Data sharing will adhere to ethical guidelines and those set by the Tiny Blue Dot Foundation, with only de-identified and aggregated data shared in accordance with FAIR principles. Sharing of data collected as part of the EAR/ Voicediary procedures will be limited to protect subject confidentiality, because raw speech data are inherently identifiable and classified as Protected Health Information (PHI). Aggregated behavioral codings and linguistic derivates of these data will be included in data files shared in accordance with the FAIR principles, but speech data and transcripts will not be shared beyond the study team.
  All data: Following publication of primary study findings, de-identified data will be made available to qualified researchers in a way that protects subject confidentiality and adheres to HIPAA policies. Informed consent documents will provide sufficient detail about the intent to archive, share, and re-analyze data.